CLINICAL TRIAL: NCT06163066
Title: The Effect of Newborn Basic Care Training Delivered With Different Methods on Fathers' Self-Efficacy and Father-Baby Attachment
Brief Title: Newborn Basic Care Training on Fathers' Self-Efficacy and Father-Baby Attachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Sevilay Ergun Arslanli, Lecturer (PhD), Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Sevilay ERGUN ARSLANLI
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Newborn Basic Care Training
Keywords: Fathers; Self-efficacy; Newborn care; Attachment; Nursing

STUDY DESIGN:
Intervention Model Description: This study will be conducted in a prospective pretest-posttest (first and fourth months) three-arm (1:1:1), randomized controlled experimental design.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Web-based Group (Experimental): The father's phone will be stolen and the father will record the researcher's phone number. After this stage, the researcher will apply a pre-test, make the father a member of the website and show the first video about basic newborn care to the father via his phone. The first access to the website will be made under the guidance of the researcher. For membership, individuals must have an internet connection and know how to use a phone. Even though the fathers made their first viewing before being discharged from the hospital, the web page will be open for 1 month and they will be able to watch the video they want whenever they want. Individuals who visit the page and agree to participate in the study will be given a posttest at the end of the 1st month and at the end of the 4th month.
  Interventions: Other: Newborn Basic Care Training
- Face-to-face Group (Experimental): The father's phone will be stolen and the father will record the researcher's phone number. Then, before his wife is discharged from the hospital, the father will be interviewed and an appointment will be made to meet at the clinic at a convenient time. During this appointment, the researcher will apply a pre-test and explain information about basic newborn care (hygiene, safety and nutrition) face-to-face and in practice. In addition, brochures about baby care will be provided to fathers that they can use at any time. After this process, the final test will be applied at the end of the 1st month and at the end of the 4th month.
  Interventions: Other: Newborn Basic Care Training
- Control Group (No Intervention): The father's phone will be stolen and the father will record the researcher's phone number. After this stage, the researcher will perform a pre-test before the mother is discharged and will not have her perform any newborn care procedures. Fathers in the control group will continue to receive routine care. In Turkey, information about the basic care of the newborn is given only verbally by neonatal midwives and nurses before discharge. After these procedures, a final test will be applied to this group at the end of the 1st month and at the end of the 4th month.

INTERVENTIONS:
Other: Newborn Basic Care Training — These talented fathers will be given both face-to-face practical training and the industrial web-based training type of information technologies will be used. In this way, the positive developments provided by the two trainings will be abandoned and the understandability and usefulness of the training from the people's perspective will be increased. A website suitable for mobile phones will be designed by transferring digital materials. With this website, fathers will be able to access information about basic care via phone whenever and wherever they want. Thus, in a short time, without human resources and time, all the fathers in need throughout the country will reach the capacity to obtain appropriate information.
  Arms: Face-to-face Group; Web-based Group

SUMMARY:
This study is planned to be carried out in a pre-test-post-test (first and fourth months) randomized controlled experimental design with the aim of determining the "Effect of Newborn Basic Care Training Given to Fathers with Different Methods on Fathers' Self-Efficacy and Father-Infant Attachment". In addition, the training provided aims to prevent malpractices in newborn care and to reduce neonatal morbidity and mortality rates and gender-based inequalities.

DETAILED DESCRIPTION:
This study will be conducted in a prospective pre-test-post-test- (first and fourth months), three-arm (1:1:1), randomized controlled experimental design.The sample size of the study was calculated based on a 3-group study on father-infant attachment. Thus, it was planned to conduct research with 73 fathers in total (24 fathers in the web-based group, 24 in the face-to-face group, and 25 in the control group).

ELIGIBILITY:
Inclusion Criteria Eligible participants were fathers who met the following criteria: (1) their spouse had given birth for the first time, (2) they were aged 18 to 50 years, (3) they consented to participate in the study and signed an informed consent form, (4) their infant was in the neonatal period, (5) they had access to a mobile phone with internet connectivity and were able to operate it, (6) they were able to read and understand xxx, (7) they had a stable living environment, (8) their child and spouse were in good health, and (9) they had no communication or visual impairments.

Exclusion Criteria:

Fathers who participated in the study but withdrew at any point, whose child or spouse experienced health complications after childbirth, or who failed to access the website within one month or engage with the educational materials, were excluded from the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — When the literature is examined, it is seen that there are a limited number of studies investigating fathers' participation in baby care and postnatal father-infant attachment. There is no study in the literature that specifically addresses the self-efficacy of fathers who are expecting their first baby or have a newborn baby, regarding the basic care of the newborn. For this reason, this study will be conducted to determine "the effect of newborn basic care training given with different methods on fathers' self-efficacy in care and father-infant attachment".
Enrollment: 73 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Fathers' Self-Efficacy Scale for Newborn Care | Change from within the first 24 hours of postpartum, after Newborn basic care training is completed (first month and fourth months) after Newborn basic care training is completed
  This scale, developed by researchers, consists of 3 sub-dimensions (Hygiene, Safety and Nutrition). The hygiene sub-dimension consists of 10 items, the security sub-dimension consists of 4 items, and the nutrition sub-dimension consists of 3 items, making a total of 17 items. Each item of the scale is scored from 1 to 5, and the lowest score obtained from the scale is 17 and the highest score is 85. A high score means that the father's self-efficacy in basic newborn care is high.
Postnatal Paternal-Infant Attachment Scale | Change from within the first 24 hours of postpartum, after Newborn basic care training is completed (first month and fourth months) after Newborn basic care training is completed
  The Postnatal Paternal-infant attachment scale is a scale developed by Condon et al. (2008) to evaluate postnatal paternal-infant attachment after birth (Condon et al., 2008). This scale was adapted to Turkish society by Güleç and Kavlak (2013) and its validity and reliability were tested. The scale consists of 3 sub-dimensions and 19 items. Each item of the scale is scored from 1 to 5, and the lowest score obtained from the scale is 19 and the highest score is 95. A high score means that attachment is high.

CONTACTS AND LOCATIONS:
Overall Officials: Sevilay ERGUN ARSLANLI, Phd Candidate, Study Director — Çankırı Karatekin University
Locations (1):
- Çankırı Karatekin University, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No